CLINICAL TRIAL: NCT03994822
Title: pRESET for Occlusive Stroke Treatment
Acronym: PROST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: phenox Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: pCT-001-19
Record Dates: First submitted 2019-05-24; First posted 2019-06-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-02

CONDITIONS: Brain Diseases; Cardiovascular Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Ischemia; Nervous System Diseases; Pathologic Processes; Stroke, Ischemic; Stroke, Acute; Vascular Diseases
Keywords: Brain; Brain Clot; Brain Infarction; Cerebral Ischemia; Cerebrovascular Disorders; Ischemia; Ischemic; Ischemic Stroke; Mechanical Thrombectomy; Neurovascular Intervention; phenox; pRESET; pRESET Thrombectomy Device; Revascularization; Randomized Control; Solitaire; Stent Retriever; Stroke; Vascular Diseases
MeSH Terms: conditions — Brain Diseases; Cardiovascular Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Ischemia; Nervous System Diseases; Pathologic Processes; Ischemic Stroke; Stroke; Vascular Diseases; Brain Infarction; Brain Ischemia

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center randomized
Who Masked: Outcomes Assessor
Masking Description: The blinded assessor performs all study assessments during and after hospital discharge (i.e., 24 hours, Day 7/Discharge (whichever is earlier), and 30 and day 90 visits
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- pRESET Thrombectomy Device (Experimental): Mechanical Thrombectomy using the pRESET Thrombectomy Device
  Interventions: Device: Mechanical Thrombectomy using the pRESET Thrombectomy device
- Solitaire Revascularization Device (Active Comparator): Mechanical Thrombectomy using the Solitaire Revascularization Device
  Interventions: Device: Mechanical Thrombectomy using the Solitaire Revascularization Device

INTERVENTIONS:
Device: Mechanical Thrombectomy using the pRESET Thrombectomy device — Clot removal using the pRESET Thrombectomy device
  Arms: pRESET Thrombectomy Device
Device: Mechanical Thrombectomy using the Solitaire Revascularization Device — Clot removal using the Solitaire Revascularization Device
  Arms: Solitaire Revascularization Device

SUMMARY:
Compare the safety and effectiveness of pRESET to Solitaire in the treatment of stroke related to large vessel occlusion

DETAILED DESCRIPTION:
To determine the safety and effectiveness of pRESET for the treatment of acute ischemic stroke within 8 hours of symptom onset (defined as time patient was last seen well) due to large vessel occlusion and to compare safety and effectiveness to the predicate device, Solitaire™ Platinum revascularization device

ELIGIBILITY:
Inclusion Criteria:

1. Age >/=18
2. Clinical signs consistent with acute ischemic stroke
3. Subject is able to be treated within 8 hours of stroke symptom onset and within 1.5 hours (90 min) from screening CT / MRI to groin puncture.
4. Pre-stroke modified Rankin Score of 0 or 1
5. NIHSS ≥6 at the time of enrolment
6. If tPA is indicated, initiation of IV tPA should be administered as soon as possible and no later than 3.0 hours of onset of stroke symptoms (onset time is defined as the last time when the patient was witnessed to be at baseline neurologic status), with investigator verification that the subject has received/is receiving the correct IV tPA dose (0.9mg/kg) for the estimated weight.
7. Expanded Thrombolysis in Cerebral Infarction (eTICI) 0-1 flow confirmed by angiography that is accessible to the mechanical thrombectomy device in the following locations:

   1. Intracranial internal carotid
   2. M1 and/or M2 segment of the MCA
   3. Carotid terminus
   4. Vertebral artery
   5. Basilar artery

   Note: M1 segment of the MCA is defined as the arterial trunk from its origin at the ICA to the first bifurcation or trifurcation into major branches neglecting the small temporo-polar branch.
8. Imaging scores as follows:

   · ASPECTS score must be 6-10 on NCCT or DWI-MRI.

   If automated core volume assessment software is used:
   * MR diffusion-weighted imaging (DWI) ≤50cc
   * Computed tomography perfusion (CTP) core ≤50 cc
9. Subject is willing to conduct protocol-required follow-up visits.
10. A valid completed informed consent by participant or LAR (Legally Authorized Representative)

Exclusion Criteria:

1. Subject who has received IA-tPA prior to enrolment in the study
2. Female who is pregnant or lactating or has a positive pregnancy test at time of admission.
3. Rapid neurological improvement prior to study enrolment suggesting resolution of signs/symptoms of stroke
4. Known serious sensitivity to radiographic contrast agents
5. Known sensitivity to nickel, titanium metals, or their alloys
6. Subjects already enrolled in other investigational studies that would interfere with study endpoints
7. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency. (A subject without history or suspicion of coagulopathy does not require INR or prothrombin time lab results to be available prior to enrolment.)
8. Known renal failure as defined by a serum creatinine > 2.0 mg/dl (or 176.8 μmol/l) or glomerular filtration rate (GFR) < 30.
9. Subject who requires hemodialysis or peritoneal dialysis, or who has a contraindication to an angiogram for whatever reason.
10. Life expectancy of less than 90 days
11. Clinical presentation suggests a subarachnoid hemorrhage, even if initial CT or MRI scan is normal
12. Suspicion of aortic dissection
13. Subject with a comorbid disease or condition that would confound the neurological and functional evaluations or compromise survival or ability to complete follow-up assessments.
14. Subject is known to currently use or has a recent history of illicit drug(s) or abuses alcohol (defined as regular or daily consumption of more than four alcoholic drinks per day).
15. Known arterial condition (e.g., proximal vessel stenosis or pre-existing stent) that would prevent the device from reaching the target vessel and/or preclude safe recovery of the device
16. Subject who requires balloon angioplasty or stenting of the carotid artery at the time of the index procedure
17. Angiographic evidence of carotid dissection

    Imaging exclusion criteria:
18. CT or MRI evidence of hemorrhage on presentation
19. CT or MRI evidence of mass effect or intra-cranial tumor (except small meningioma)
20. CT or MRI evidence of cerebral vasculitis
21. CT or MRI-DWI showing ASPECTS 0-5. Alternatively, if automated core volume assessment software is used, MRI-DWI or CTP core > 50cc.
22. CT/MRI shows evidence of carotid dissection or complete cervical carotid occlusion requiring a stent
23. Any imaging evidence that suggests, in the opinion of the investigator, the subject is not appropriate for mechanical thrombectomy intervention (e.g. inability to navigate to target lesion, moderate/large infarct with poor collateral circulation, etc.).
24. Occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation) as confirmed by angiography, or clinical evidence of bilateral strokes or strokes in multiple territories

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-05-12 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: Patients with a Modified Rankin Scale (mRS) </= 2 | 90 (+/-15) days
  Global disability assessed via the blinded evaluation of the proportion of patients with a Modified Rankin Scale (mRS) </= 2
Primary Safety Endpoint: Device- or procedure-related symptomatic intracerebral hemorrhage (sICH) | 24 (-8/+12) hours
  Proportion of subjects with device- or procedure-related symptomatic intracerebral hemorrhage (sICH)

SECONDARY OUTCOMES:
Successful Revascularization measured using the expanded Thrombolysis in Cerebrovascular Infarction (eTICI) | During Index Procedure
  Proportion of subjects with eTICI 2b50 or greater flow in the target vessel post procedure with 3 or fewer passes of the assigned study device.
Successful Revascularization on first pass measured using the expanded Thrombolysis in Cerebrovascular Infarction (eTICI) | During Index Procedure
  Proportion of patients with eTICI 2c or greater, following the first pass of the assigned study device
Overall mortality following the index stroke | 90 (+/-15) days
  Overall mortality following the index stroke
Distribution of mRS shift across the entire spectrum of disability | 90 (+/-15) days
  Distribution of mRS shift across the entire spectrum of disability

CONTACTS AND LOCATIONS:
Overall Officials: Raul G Nogueira, MD, Principal Investigator — University of Pittsburgh Medical Center, Pittsburgh; Richardo A Hanel, MD, Principal Investigator — Baptist Medical Center Jacksonville
Locations (24):
- United States (19):
  - Honor Health Research Institute, Scottsdale, Arizona
  - Providence Little Company of Mary Medical Center, Santa Monica, California
  - University of Miami, Coral Gables, Florida
  - Baptist Health Research Institute Jacksonville, Jacksonville, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Advocate Lutheran General Hospital, Downers Grove, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Massachusetts, Worcester, Massachusetts
  - JFK Medical Center, Edison, New Jersey
  - Buffalo General Medical Center, Buffalo, New York
  - NYU Langone Health, New York, New York
  - The Mount Sinai Hosptial, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - OhioHealth Research Institute, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - Valley Baptist, Harlingen, Texas
  - Swedish Medical Center - Cherry Hill Campus, Seattle, Washington
- Germany (5):
  - Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum rechts der Isar Technische Universität München, München, Bavaria
  - Klinikum Bremen-Mitte, Bremen, Lower Saxony
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Helios Klinikum Erfurt GmbH, Erfurt, Thuringia

IPD SHARING:
Plan to Share IPD: No